CLINICAL TRIAL: NCT01648062
Title: Using Mental Imagery to Deliver Self-Regulation Techniques That Target Sleep Initiation Behaviors and Pre-Sleep Arousal
Brief Title: Sleep Self-Regulation Using Mental Imagery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Dr Marisa Loft, Lecturer, University of Auckland, New Zealand
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IISleepTrial12
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Sleep Deprivation; Insomnia
Keywords: Sleep; self-regulation; Implementation intentions; intervention; mental simulation
MeSH Terms: conditions — Sleep Deprivation; Sleep Initiation and Maintenance Disorders; Self-Control | interventions — Imagery, Psychotherapy; Sleep; Professional Autonomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arousal reduction using guided imagery (Active Comparator): Sleep Self-Regulation Using Mental Imagery: Participants in the arousal reduction condition were instructed to imagine wearing a backpack loaded with their worries, then putting the heavy backpack down, and then experiencing the relief and freedom from tension.
  Interventions: Behavioral: Sleep Self-Regulation Using Mental Imagery
- Mental simulation of sleep behavior (Active Comparator): Sleep Self-Regulation Using Mental Imagery: Participants in this condition received instructions to visualize a specific behavioral plan designed to meet the goal of obtaining quality sleep each night through the practice of certain behaviors. To form the behavioral plan, participants visualised changing into comfortable clothes and taking time to relax prior to going to bed, the time they planned to go to sleep, where they planned to sleep, and the bedtime routine they follow to help them to get to sleep. At bedtime, they were instructed to mentally run through a checklist of these behaviors and then do any behaviors that they had not yet completed.
  Interventions: Behavioral: Sleep Self-Regulation Using Mental Imagery
- Combination (Active Comparator): Sleep Self-Regulation Using Mental Imagery: Participants in this condition were asked to practice a combination of the guided imagery (for relaxation) and mental simulation imagery for sleep-related behaviour
  Interventions: Behavioral: Sleep Self-Regulation Using Mental Imagery
- Control (Sham Comparator): Sleep Self-Regulation Using Mental Imagery: Participants in this condition were asked to imagine a typical post work activity
  Interventions: Behavioral: Sleep Self-Regulation Using Mental Imagery

INTERVENTIONS:
Behavioral: Sleep Self-Regulation Using Mental Imagery — Comparison of two forms of mental imagery to instigate behaviors that assist in the sleeping process
  Other Names: mental imagery; guided imagery; Implementation intentions; sleep; self-regulation; behavior change

SUMMARY:
This randomised controlled trial assessed the efficacy of four mental imagery techniques for improving sleep and its related behaviour: (1) imagery focused on reducing arousal levels; (2) imagery incorporating implementation intentions (a strategy designed to link specified behaviour with the anticipated context) for sleep-related behaviour; (3) a combination of imagery using arousal reduction and implementation intention strategies; or (4) a condition where participants were asked to imagine their typical post work activities.

DETAILED DESCRIPTION:
Sleep deprivation is a significant health issue in the modern workplace. We conducted a randomized controlled trial to test the efficacy of techniques involving mental imagery promoting relaxation (arousal reduction; AR) and simulation of the appropriate sleep behavior in the likely environments (implementation intentions; II) in a population of daytime employees

ELIGIBILITY:
Inclusion Criteria:

* ability to read and write in English;
* full-time employment;
* work shifts during daytime hours (i.e., participants were excluded if they worked night shifts either through the organization or through a secondary job) in a position that provided daily access to email;
* a score of five or greater on the Pittsburgh Sleep Quality Inventory (PSQI) which indicates at least moderate difficulties in two or more areas (e.g., sleep quality and daytime dysfunction);

Exclusion Criteria:

* An identifiable biological cause of current sleep deprivation (e.g., sleep apnoea, narcolepsy, restless leg syndrome, periodic limb movement disorder, or pregnancy)
* An identified psychological disorder
* Caring for a child under the age of 5 or have a reason outside of work that caused them to regularly lack sleep.
* Incomplete data (over 50% of daily data missing or missing final follow-up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Baseline and at 3 weeks. Data will also be presented for every day for the duration of the 3 week period so change can be reported.
  Assessed using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al, 1989).The PSQI includes 19 items that assess sleep quality, hours of sleep, sleep onset length, sleep efficiency, sleep disturbances, use of medication and daytime. Item ratings are recoded and combined to form seven component scores. These scores are then summed into a global score ranging from 0(no difficulty) to 21(severe difficulties in all areas). Daily sleep quality was assessed with five PSQI items.

SECONDARY OUTCOMES:
Negative Sleep Habits | Baseline and Final follow-up (at 21-days)
  The Sleep Hygiene Index (Mastin et al, 2006). Respondents rate on a scale from 1 (never) to 5 (all the time) how frequently they engaged in 13 behaviors (e.g. "I take naps lasting two or more hours"). Ratings were summed to provide a total negative sleep habit frequency score.
Sleep Efficacy | Baseline and final follow-up (at 21 days)
  Participants rated their sleep self-efficacy with the item, "how confident are you that you can take the actions necessary to get a good sleep tonight?" Sleep response efficacy was rated with the item "how confident are you that you will actually get a good sleep tonight?" ratings ranged from 1 (not at all confident) to 10 (very confident), and they were summed; r=.69, p<.01 at baseline and r=.20, p<.05 at final follow-up.
Pre-Sleep Arousal | Baseline and final follow-up (Day 21)
  The Pre-sleep Arousal Scale (Nicasso et al, 1985) includes an 8-item somatic subscale (e.g. "how often in the last week before bed have you had a tight, tense feeling in your muscles?") and an 8-item cognitive subscale (e.g. "how often in the last week before bed do you review or ponder events of the day?"). Ratings range from 1 (not at all) to 5 (extremely) and are summed to generate scores.
Imagery Adherence | Post-session, Daily, Final follow-up (21 days)
  Measure adapted from the Vividness of Imagery Questionnaire (White et al, 1978). Participants rated the vividness of the following images: (1) putting things into a bag, (2) releasing a bag, (3) getting home from work, (4) relaxing at home, (5) their night-time routine, (6) the time that they visualised going to bed, (7) the environment of their bedroom, (8) the details of the bed they are sleeping in, (9) the image of themselves falling asleep. Response options were: 1 (no image at all) 2 (vague and dim), 3 (somewhat vivid), 4 (reasonably clear), and 5 (perfectly clear and vivid).
Action Planning | Baseline, Final follow-up (Day 21)
  An adaptation of the action planning measure developed by Luszczynska and Schwarzer (2003) was used. The items included: "I have made a detailed plan for (1) how I am going to wind down before going to sleep (2) how I am going to prepare for bed (3) how I am going to prepare the place where I will sleep, and (4) the time when I go to sleep". Responses ranged from 1 (not at all) to 7 (very much); ratings were summed to generate scores.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa H Loft, PhD, Principal Investigator — Monash University (Sunway Campus, Malaysia); Linda D Cameron, PhD, Study Director — University of California, Merced
Locations (1):
- 10 Private Businesses in the Region, Auckland, New Zealand